CLINICAL TRIAL: NCT06750835
Title: Efficacy of the Serratus Posterior Superior Intercostal Plane Block for Postoperative Analgesia in Breast Cancer Surgery : A Randomized Comparative Study
Brief Title: Efficacy of the Serratus Posterior Superior Intercostal Plane Block for Postoperative Analgesia in Breast Cancer Surger.(SPSIP) Block is a Novel Regional Anesthesia Technique Targeting the Dorsal Rami and Intercostal Nerves (T2-T6), Providing Sensory Blockade to Both the Posterior and Lateral Aspect
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rehab Adel Ebrahim Okely (Other)
Responsible Party: Sponsor-Investigator, Rehab Adel Ebrahim Okely, Assistant lecturer, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPSIP block in breast cancer
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SPSIP block (Active Comparator): Serratus posterior superior intercostal plane block
  Interventions: Procedure: SPSIP block
- SAP block (Active Comparator): Serratus anterior plane block
  Interventions: Procedure: SAP block
- Paravertebral block (Active Comparator): Paravertebral block
  Interventions: Procedure: Paravertebral block

INTERVENTIONS:
Procedure: SPSIP block — Serratus posterior superior intercostal plane block
  Arms: SPSIP block
Procedure: SAP block — Serratus anterior plane block
  Arms: SAP block
Procedure: Paravertebral block — * The block will be administered under ultrasound guidance at the T2-T5 levels.
  * A total of 15 mL of 0.25% bupivacaine will be injected into the paravertebral space on the side of the surgery.
  Arms: Paravertebral block

SUMMARY:
The Serratus Posterior Superior Intercostal Plane (SPSIP) block is a novel regional anesthesia technique targeting the dorsal rami and intercostal nerves (T2-T6), providing sensory blockade to both the posterior and lateral aspects of the chest wall. By blocking these nerves at a more posterior location, the SPSIP block can potentially offer broader and more comprehensive analgesia for breast surgeries, including the axillary and deeper structures of the breast. This makes it a promising alternative or adjunct to the existing regional techniques used in breast cancer surgeries

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy among women worldwide, often requiring surgical intervention such as mastectomy or breast-conserving surgery. Despite advancements in surgical techniques, postoperative pain remains a significant concern, as inadequate pain management can lead to delayed recovery, increased opioid consumption, and a higher incidence of chronic pain conditions such as postmastectomy pain syndrome (PMPS). Effective pain control strategies are, therefore, crucial to enhancing patient recovery, reducing hospital stay, and improving overall quality of life [1].

Regional anesthesia techniques have gained prominence as an effective method for perioperative pain management in breast surgery [2]. Traditional blocks such as the Thoracic Paravertebral Block (TPVB) and Serratus Anterior Plane (SAP) Block have been extensively studied and are considered effective options for postoperative analgesia. However, these techniques are not without limitations [3]. The TPVB, although effective, carries a higher risk of complications such as pneumothorax and hypotension due to its proximity to the pleura. The SAP block, on the other hand, primarily provides analgesia to the lateral thoracic wall and may not adequately cover deeper breast tissues and posterior thoracic areas The current study aims to evaluate the efficacy of the SPSIP block for postoperative analgesia in breast cancer surgeries and to compare its analgesic profile with the SAP block and TPVB. By providing a comprehensive comparison, this study seeks to establish the SPSIP block as a viable and potentially superior option for postoperative pain management in breast cancer surgery.

> Patients and methods

• Type of the Study: This is a prospective, randomized controlled cohort study comparing the efficacy of the Serratus Posterior Superior Intercostal Plane (SPSIP) Block, Serratus Anterior Plane (SAP) Block, and Thoracic Paravertebral Block (PVB) for postoperative analgesia in breast cancer surgery.

• Study Setting: The study will be conducted at Assiut University Hospital, a tertiary care center equipped with advanced facilities for breast cancer surgeries and postoperative pain management.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18-75 years. 2. Scheduled for elective breast cancer surgery (MRM or BCS). 3. ASA physical status I-II. 4. Able to provide written informed consent.

-

Exclusion Criteria:

1. Chronic pain conditions or long-term opioid use. 2. Coagulation disorders (platelets < 100,000/mm³ or INR > 1.5). 3. Severe obesity (BMI > 35 kg/m²). 4. Allergy to local anesthetics. 5. Anatomical abnormalities affecting block placement. 6. Pregnant or lactating women. 7. Active infection or skin lesions at the injection site.

-

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Post operative pain relief | 24 hours
  the level of postoperative pain as assessed by the Numerical Rating Scale (NRS) at rest and during movement at predefined intervals: 1 hour, 6 hours, 12 hours, and 24 hours post-surgery. The NRS is a validated tool that ranges from 0 (no pain) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
Total Opioid Consumption | 24 hours
Time to First Analgesic Request | 24 hours
Incidence of Postoperative Nausea and Vomiting (PONV) | 24 hours